CLINICAL TRIAL: NCT00887172
Title: A Randomized Double Blind, Placebo-Controlled Clinical Trial of Chinese Herbal Medicine (CHM) in the Treatment of Acute Upper Respiratory Tract Infections
Brief Title: Trial of Chinese Herbal Medicine in the Treatment of Upper Respiratory Tract Infections (URTIs)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Research Fund for the Control of Infectious Diseases of the Food and Health Bureau, the Government of the Hong Kong SAR (Unknown)
Responsible Party: Cindy L. K. Lam, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKCTR-6
Record Dates: First submitted 2009-04-06; First posted 2009-04-23 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Acute Upper Respiratory Tract Infections
Keywords: Acute upper respiratory tract infections
MeSH Terms: interventions — jing fang bai du san

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Wind-cold syndrome group were patients classified by Chinese Medicine practitioner of Wind-cold syndrome and took treatment of Jing Fang Bai Du san.
  Interventions: Drug: Jing Fang Bai Du san
- 2 (Placebo Comparator): Wind-cold syndrome group were patients classified by Chinese Medicine practitioner of Wind-cold syndrome and took placebo of Jing Fang Bai Du san.
  Interventions: Drug: Placebo
- 3 (Experimental): Wind-heat syndrome group were patients classified by Chinese Medicine practitioner of Wind-heat syndrome and took treatment of Ying Qiao san.
  Interventions: Drug: Ying Qiao san
- 4 (Placebo Comparator): Wind-heat syndrome group were patients classified by Chinese Medicine practitioner of Wind-heat syndrome and took placebo of Ying Qiao san.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jing Fang Bai Du san — The Jing Fang Bai Du san can relieve external symptoms and effectively clear up the pathogenic cold. It contains 13 herbs including, Radix Angelicae Pubescentis, Radix Peucedani, Radix Ginseng, Smilacis Glabrae Rhizoma, Rhizoma Chuanxiong, Fructus Aurantii, Radix Platycodi, GlycyrrhizaeRadix, Herba Schizonepetae, Fructus Arctii, MenthaeFolium, Radix Saposhnikoviae, Rhizoma et Radix Notopterygii.The CHM preparations were manufactured and supplied by Pura Pharm International (H.K.) Ltd., in the form of concentrated granules which follows the GMP standard. None of the herbs in these two formulas are included in the Toxic Chinese Herbal Medicine List of the Chinese Medicine Ordinance Schedule 1 or being a controlled substance, animal product, or endangered species.
  Arms: 1
Drug: Placebo — The sachets of the CHM formulae and placebo were identical in appearance except for the randomization numbers. The placebo contains Maltose-dextrine granules that are identical in weight, appearance, flavour and texture as the CHM granules. Both the Chinese medicine practitioner who assessed the subjects and the subjects were blinded to the nature of the treatment. The pharmaceutical supplier kept the medication and placebo codes, which were broken at the end of the study after completion of all the assessment and data analyses.
  Arms: 2; 4
Drug: Ying Qiao san — The Ying Qiao san can relieve external symptoms and effectively clear up the pathogenic heat. It contains 10 herbs: Fructus Forsythiae, LoniceraeFlos, Radix Platycodi, MenthaeFolium, GlycyrrhizaeRadix, Herba Schizonepetae, Sojae Semen praeparatum, Fructus Arctii, PhragmitisRhizoma and LophatheriHerba. The CHM preparations were manufactured and supplied by Pura Pharm International (H.K.) Ltd., in the form of concentrated granules which follows the GMP standard. None of the herbs in these two formulas are included in the Toxic Chinese Herbal Medicine List of the Chinese Medicine Ordinance Schedule 1 or being a controlled substance, animal product, or endangered species.
  Arms: 3

SUMMARY:
Upper respiratory tract infections (URTIs) are the most common illnesses in primary medical services but there is no established cure for these conditions in Western medicine. In Hong Kong, many patients use Chinese herbal medicine (CHM) for the treatment of URTIs but there is little research evidence on their effectiveness or side effects. The aim of this study is to test whether two commonly used Chinese herbal medicine (CHM) formulae guided by Traditional Chinese medicine (TCM) diagnosis will significantly increase recovery rate, and reduce the duration and/or severity of symptoms, and improve the quality of life of patients with URTIs in primary care.

If a patient consents to take part in the study and is found eligible, he/she will be invited by the consulting doctor, and then be assessed by a registered Chinese medicine practitioner for whether the illness satisfies the TCM diagnosis of the two major TCM types of URTIs: Group A (Wind-cold syndrome) and Group B (Wind-heat syndrome). Subjects in Group A (Wind-cold syndrome) will be randomised to receive the Jing Fan Bai Du san or placebo. Subjects in Group B (Wind-heat syndrome) will be randomised to receive Ying Qiao san or placebo. Both group A and B treatments and placebo will be given in sachets of granules that are identical in appearance. Neither the Chinese medicine practitioner, the recruiting doctors, nor patient know whether a subject is taking CHM or placebo.

328 subjects (164 in each diagnosis group) will be recruited from patients consulting the Ap Lei Chau Government General Outpatient clinic for URTIs. Each subject is required to return to the clinic for follow-up assessment by the Chinese medicine practitioner on day 7 post-treatment and all subjects will be contacted by telephone on Day 2, 3, 5, 9, 11, 13,15 and 20 after treatment to assess their symptoms and to find out if they have developed any side effects or adverse reactions.

The main outcome measure is any difference in the proportion of subjects who have resolution of the URTI on Day 7 between the treatment and placebo groups. The secondary outcome measures are the reduction in the duration and severity of symptoms, quality of life during the illness and side effects.

This study will provide scientific evidence to support or refute the effectiveness of two commonly used CHM formulae in the treatment of URTIs.

DETAILED DESCRIPTION:
Acute upper respiratory tract infections (URTIs) are the most common diagnoses made in the primary medical services, which consisted of 34.6% of all diagnoses in Hong Kong. It accounts for approximately 100 million visits per year in the US. It was estimated that an adult has an average of 3 to 4 times while children has an average of 6 to 8 times each year. WHO has pointed out that URTIs have a great impact on personal and economical aspects although they are rarely lethal It was estimated that 60% of the working class has contracted URTIs each year, and a loss of 8.8 days of perfect health for each worker on average each year, and a loss of up to HK$ 31.3 billion of economic output each year.

There is no established curative treatment in Western medicine for URTIs except for selected cases of influenza. Studies have shown that the average duration of illness of an URTI is around 7 days, and most URTIs resolve by the 10th day. Traditional Chinese medicine (TCM) is commonly used by people in Hong Kong on its own or along side with Western medicine for the treatment of URTIs. The Chinese Medicine Council of Hong Kong was established in September 1999, the use of Chinese herbal medicine (CHM) is expected to increase and there is an urgent need for research evidence on their effectiveness and side effects. TCM follows a theoretical and methodological pathway, which leads to its diagnosis and treatment. Most URTIs can be differentiated into two types according to the theory of TCM: Wind-cold syndrome and Wind-heat syndrome. The theory leads to two classical herbal formulae that are very popular in Hong Kong: the Jing Fang Bai Du san for treating the Wind-cold syndrome whiles the Ying Qiao san for treating Wind-heat syndrome.

The Jing Fang Bai Du san can relieve external symptoms and effectively clear up the pathogenic cold. It contains 13 herbs including, Radix Angelicae Pubescentis, Radix Peucedani, Radix Ginseng, Smilacis Glabrae Rhizoma, Rhizoma Chuanxiong, Fructus Aurantii, Radix Platycodi, GlycyrrhizaeRadix, Herba Schizonepetae, Fructus Arctii, MenthaeFolium, Radix Saposhnikoviae, Rhizoma et Radix Notopterygii. Previous clinical studies conducted in China showed mixed results on the effectiveness of Jing Fang Bai Du san on Wind-cold syndrome. One study showed that it was no better than no treatment while another study showed that concentrated granules of Jing Fang Bai Du san was more effective (80%) than Western medicine (10%) in improving and resolving symptoms of Wind-cold syndrome within 7 days.

The Ying Qiao san can relieve external symptoms and effectively clear up the pathogenic heat. It contains 10 herbs: Fructus Forsythiae, LoniceraeFlos, Radix Platycodi, MenthaeFolium, GlycyrrhizaeRadix, Herba Schizonepetae, Sojae Semen praeparatum, Fructus Arctii, PhragmitisRhizoma and LophatheriHerba. From pharmacological studies, it showed anti-inflammatory, antipyretic, analgesic, anti-bacterial and antiviral actions. A clinical trial also showed the concentrated granules of Ying Qiao san was more effective (66.13%) than Western medicine (40%) in resolving the symptoms of Wind-heat syndrome within 1 week. These two CHM formulae have been used for many years and have not been associated with any serious adverse reactions. The common side effects are mild diarrhoea and headache.

Although there are some data from Mainland China suggesting the effectiveness of these two formulae for URTIs but most of these previous studies were observational and the few clinical trials were not placebo-controlled and of poor quality. Furthermore, results of trials from Mainland China may not be generalisable to the people in Hong Kong. Most previous studies on CHM focused on individual herbs, which is against the TCM principles as pointed out by the WHO. The WHO recommends that future clinical studies should attempt to integrate TCM diagnosis pattern with traditional CHM treatments. In this proposed study, the integrated TCM approach of using traditional formulae of multiple herbs, guided by the TCM diagnosis, will be used in a double-blind randomized placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they have all the following:

  * Age ≥18 years old
  * Patient has developed URTIs symptoms for 48 hours or less.
  * At least one from each of the following groups of URTIs symptoms:
* Symptoms of infection: headache, chills, muscle ache, or an oral temperature greater than 37.5 degrees Celsius.
* Symptoms from the upper respiratory tract: cough, hoarseness, running nose, nasal obstruction, itchy throat, sore throat or sneezing.

Exclusion Criteria:

* Patients will be excluded from the study if they have one or more of the following:

  * Have symptoms of URTIs for more than 48 hours.
  * Pregnancy or breast-feeding
  * Liver disease
  * Known immune deficiency
  * Alcohol (>30 units/wk) or drug abuse
  * Medical history of asthma, allergic rhinitis, cystic fibrosis and chronic bronchopulmonary diseases
  * Known allergies to food additives or study medications
  * Taking chronic medications that contain any kind of herbs, mineral, or specific vitamin supplements
  * Diabetes mellitus
  * Cancer
  * Any other serious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the proportion of patients who will have resolution on day 7. | day 7

SECONDARY OUTCOMES:
The secondary outcome measures are the duration from onset of the illness to the resolution of symptoms, change in daily symptom scores, SF-36 health-related quality of life scores and side effects. | on day 0, 1, 4, 7, 10, 14, 20 and 21

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L K Lam, MD, Principal Investigator — Family Medicine Unit, Faculty of Medicine, HKU
Locations (1):
- Two General Outpatient Clinics, Hong Kong, Hong Kong, China